CLINICAL TRIAL: NCT00603642
Title: A Randomized, Double Blind, Placebo Controlled Phase 3 Study Evaluating the Efficacy and Safety of AMG 531 in Thrombocytopenic Japanese Subjects With Immune (Idiopathic) Thrombocytopenic Purpura
Brief Title: P3 Study to Evaluate Efficacy and Safety of AMG 531 in Thrombocytopenic Japanese Subjects With Immune (Idiopathic) Thrombocytopenic Purpura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060216
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: AMG 531; Idiopathic Thrombocytopenic Purpura; ITP; Thrombocytopenia; Japan; Placebo controlled; Phase 3
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 531 (Placebo Comparator): Double blinded placebo-controlled study
  Interventions: Drug: AMG 531
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subcutaneously administered, once a week, for 12 weeks
  Arms: Placebo
Drug: AMG 531 — Subcutaneously administered, once a week, for 12 weeks
  Arms: AMG 531

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AMG 531 compared with placebo in thrombocytopenic Japanese subjects with immune (idiopathic) thrombocytopenic purpura (ITP) .

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with diagnosis of ITP according to the diagnostic criteria proposed by Research Committee for Idiopathic Hematopoietic Disorders of the Ministry of Health, Labour and Welfare [MHLW] (revised in 1990) at least 6 months before the first screening visit
* The mean of the 3 scheduled platelet counts taken at the scheduled visits during the screening period must be ≤ 30 x 10^9/L, with no individual count > 35 x 10^9/L
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Subjects must be ≥ 20 years of age at the time of obtaining the informed consent
* Have received at least 1 prior treatment for ITP
* If known Helicobacter pylori positive, having completed one course of Helicobacter pylori eradication therapy at least 12 weeks before the first screening visit
* A hemoglobin value taken at scheduled visit during the screening period must be ≥ 10 g/dL
* A serum creatinine concentration taken at scheduled visit during the screening period must be ≤ 2 mg/dL
* Adequate liver function, as evidenced by a total bilirubin taken at scheduled visit during the screening period ≤ 1.5 times of the upper limit of the normal range (except for patients with a confirmed diagnosis of Gilbert's Disease) or an alanine aminotransferase and aspartate aminotransferase taken at the screening visit ≤ 3 times of the upper limit of the normal range

Exclusion Criteria:

* Any known history of bone marrow stem cell disorder. Any abnormal bone marrow findings other than those typical of ITP.
* Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, no treatment or active disease within 5 years before the first screening visit.
* Documented diagnosis of arterial thrombosis (eg, stroke, transient ischemic attack, or myocardial infarction); history of venous thrombosis (eg, deep vein thrombosis, pulmonary embolism) and receiving anticoagulation therapy at the first screening visit.
* Documented diagnosis of anti phospholipid antibody syndrome
* Currently receiving any treatment for ITP except oral corticosteroids, azathioprine and/or danazol administered at a constant dose and schedule from at least 4 weeks prior to the first screening visit
* Received intravenous immunoglobulin, anti D immunoglobulin, or any drug administered to increase platelet counts (eg, immunosuppressants except azathioprine) within 2 weeks before the first screening visit
* Have had a splenectomy for any reason within 12 weeks before the first screening visit
* Past or present participation in any study evaluating pegacaristim (polyethylene glycol-conjugated recombinant human megakaryocyte growth and development factor, KRN9000), Eltrombopag (SB 497115), recombinant human thrombopoietin, AMG 531, or other Mpl stimulation product
* Received hematopoietic growth factors (eg, granulocyte colony stimulating factor, macrophage colony stimulating factor, erythropoietin, interleukin 11) for any reason within 4 weeks before the first screening visit
* Received any anti malignancy agents (eg, cyclophosphamide, 6 mercaptopurine, vincristine, vinblastine, Interferon alfa) for any reason within 8 weeks before the first screening visit
* Received any monoclonal antibody drugs (eg, rituximab) for any reason within 14 weeks before the first screening visit
* Less than 4 weeks since receipt of any therapeutic drug or device that is not MHLW approved for any indication before the first screening visit
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* Known severe drug hypersensitivity
* Concerns for subject's compliance with the protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2009-04-13 (Actual); Study Completion 2009-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 20 November 2007 through 11 December 2008
Groups:
- Placebo: Placebo administered subcutaneously once weekly for 12 weeks
- Romiplostim: Romiplostim administered subcutaneously once weekly for 12 weeks at a starting dose of 3 µg/kg
Period: Overall Study
Arm/Group | Placebo | Romiplostim
Started | 12 | 22
Completed | 12 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romiplostim | Total
Number analyzed (Participants) | 12 | 22 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (13.4) | 58.5 (12.6) | 54.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 2 | 8 | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 12 | 22 | 34
  Other | 0 | 0 | 0
Platelet Count [Mean (Standard Deviation); unit: 10^9/L] | 15.8 (8.6) | 18.4 (8.3) | 17.5 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Weeks With Weekly Platelet Response
Description: Number of weeks with weekly platelet response. A weekly platelet response is defined as a platelet count of ≥ 50 x 10^9/L on a weekly scheduled dose day from week 2 to week 13.
Time Frame: 12 weeks (Weeks 2 - 13)
Population: Full Analysis Set, composed of all randomized participants who received at least 1 dose of romiplostim or placebo
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 12 | 22
Weeks | 0.0 [0.0 to 0.0] | 11.0 [9.0 to 12.0]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Increased Platelet Count From Baseline of at Least 20 x 10^9/L
Description: An increase in platelet count of at least 20 x 10^9/L from baseline within the participant during the treatment period. Increase was calculated as the maximum observed platelet count during the treatment period minus the baseline platelet count.
Time Frame: Baseline, 12 weeks (Weeks 2 - 13)
Population: Full Analysis Set, composed of all randomized participants who received at least 1 dose of romiplostim or placebo
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 12 | 22
Participants | 3 | 21
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Change From Baseline in Mean of Last 4 Weekly Platelet Counts
Description: Change from baseline in the mean of the last 4 weekly platelet counts from week 2 to week 13.
Time Frame: 12 weeks (Weeks 2 - 13)
Population: Full Analysis Set, composed of all randomized participants who received at least 1 dose of romiplostim or placebo
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 12 | 22
10^9/L | 2.3 (6.5) | 109.7 (88.5)
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.0003, ANCOVA

4. Secondary Outcome: Weeks With Platelet Count Between 50 and 200
Description: Number of weeks with platelet count between 50 x 10^9/L and 200 x 10^9/L inclusive during week 2 to week 13.
Time Frame: 12 weeks (Weeks 2 - 13)
Population: Full Analysis Set, composed of all randomized participants who received at least 1 dose of romiplostim or placebo
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 12 | 22
Weeks | 0.2 (0.4) | 6.3 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rescue Medication(s)
Description: Requirement for rescue medication(s) during treatment by the participant
Time Frame: 12 weeks (Weeks 2 - 13)
Population: Full Analysis Set, composed of all randomized participants who received at least 1 dose of romiplostim or placebo
Measure: Number; unit: Participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 12 | 22
Participants | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.6015, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12 weeks of treatment plus follow-up period up to 12 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Romiplostim
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/22
Other Adverse Events (participants affected / at risk) | 11/12 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romiplostim (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Romiplostim (N=22)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Eyelid function disorder (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Feeling abnormal (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 4
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 9
Pharyngitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
White blood cell count increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 2
Polymenorrhagia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.